CLINICAL TRIAL: NCT04121910
Title: An Open-label, 3-period Fixed-sequence Study in Healthy Subjects to Assess the Pharmacokinetics (PK) of Savolitinib When Administered Alone and in Combination With Itraconazole
Brief Title: A Study to Evaluate the Amount of Drug That Becomes Available in the Blood Circulation When Savolitinib is Administered Alone and in Combination With Itraconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: D5084C00002
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Solid Tumour
Keywords: Pharmacokinetics; Safety; Small molecule kinase inhibitor; Open-label
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Savolitinib and/or Itraconazole (Experimental): Treatment Period 1: Single administration of savolitinib (200 mg) will occur on Study Day 1 after a high-fat, high-calorie breakfast followed by PK sampling for 48 hours Treatment Period 2: Itraconazole will be administered (200 mg BID) on Study Day 15, and (200 mg QD) on Study Days 16 and 17, 1 hour before breakfast (and before dinner, when applicable) Treatment Period 3: A single combination of itraconazole (200 mg) 1 hour before breakfast + savolitinib (200 mg) after a high-fat, high-calorie breakfast on Study Day 18, and a single dose of itraconazole (200 mg) on Study Day 19, 1 hour before breakfast
  Interventions: Drug: Savolitinib; Drug: Itraconazole

INTERVENTIONS:
Drug: Savolitinib — On Study Day 1 and Study Day 18, savolitinib will be administered as single dose after a high-fat, high-calorie breakfast
Drug: Itraconazole — Twice daily on first day of dosing (Study Day 15) followed by once daily for 4 days (Study Day 16 - Study Day 19) administered 1 hour before any breakfast (and 1 hour before dinner on Study Day 15)

SUMMARY:
This study will be conducted to quantify the magnitude of the effect of itraconazole co-administration on the PK of savolitinib. The exposure to savolitinib is predicted to increase when co-administered with the potent cytochrome P (CYP) 3A4 inhibitor itraconazole since CYP3A4 (via CYP450) is involved in the metabolism and elimination of savolitinib.

DETAILED DESCRIPTION:
This study will be an open-label, 3-period, fixed-sequence study in non-Japanese healthy male subjects conducted at a single study centre.

The study will comprise:

1. A screening period of maximum 28 days;
2. Three treatment periods:

   1. Treatment Period 1 consists of 15 days with admission on Study Day -1, followed by a single dose administration of savolitinib on Study Day 1 followed by a washout period of at least 14 days. Subjects will be discharged from the study centre on Day 3, after the last PK sample is collected.
   2. Treatment Period 2 consists of 4 days with admission on Study Day 14, followed by itraconazole administration for 3 days (200 mg BID on Study Day 15, 200 mg QD on Study Days 16 and 17).
   3. Treatment Period 3 consists of 3 days, starting immediately after the end of Treatment Period 2 comprising of single dose administration of savolitinib (200 mg) on Study Day 18 and itraconazole administration (200 mg QD) on Study Days 18 and 19. The subjects will be discharged from the study centre on Study Day 20 after the last PK sample.
3. The Follow-up Visit will occur at least 14 days after the last dose of savolitinib PK sample in Treatment Period 3.
4. Subjects will be admitted to the study centre on 2 different occasions: Study Day-1 (Study Day -1) to Study Day 3 of Treatment Period 1 and Day -1 (Study Day 14) of Treatment Period 2 to Day 3 (Study Day 20) of Treatment Period 3.

The study drugs will be administered as follows:

1. Treatment Period 1: Single administration of savolitinib (200 mg) will occur on Study Day 1 after a high-fat, high-calorie breakfast followed by PK sampling for 48 hours.
2. Treatment Period 2: Itraconazole administered BID (200 mg BID) on Study Day 15, and (200 mg QD) on Study Days 16 and 17, 1 hour before breakfast (and before dinner, when applicable).
3. Treatment Period 3: A single combination of itraconazole (200 mg) 1 hour before breakfast + savolitinib (200 mg) after a high-fat, high-calorie breakfast on Study Day 18, and a single dose of itraconazole (200 mg) on Study Day 19, 1 hour before breakfast.

Each subject will be involved in the study for up to 60 days.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male subjects with suitable veins for cannulation or repeated venipuncture: non-Japanese male subjects aged 18 to 65 years (inclusive).
3. Have a body mass index between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
4. Alanine aminotransferase, aspartate aminotransferase and total bilirubin within normal limits for the institution at screening and Day -1.
5. Have a calculated creatinine clearance greater than 60 mL/min using the Cockcroft-Gault formula at Screening.
6. Provision of signed, written and dated informed consent for optional genetic/biomarker research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in the protocol.

Exclusion criteria:

1. Healthy subjects of Japanese ethnicity and any healthy subject that has 1 parent or grandparent (maternal or paternal) of Japanese ethnicity.
2. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
3. History or presence of GI, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
4. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
5. Planned in-patient surgery, dental procedure or hospitalisation during the study.
6. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the PI.
7. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
8. Abnormal vital signs, after 5 minutes supine rest at screening and Day -1, defined as any of the following:

(1) Systolic BP <90 mmHg or ≥140 mmHg (2) Diastolic BP <50 mmHg or ≥90 mmHg (3) Heart rate <45 or >85 beats per minute (BPM) 9) Any clinically important abnormalities in rhythm, conduction or morphology of the 12-lead resting ECG that may interfere with the interpretation of QTc interval changes.

These include healthy subjects with any of the following:

1. Abnormal ST-T-wave morphology, particularly in the protocol defined primary lead (V2) or left ventricular hypertrophy.
2. PR interval shortening <120 ms (PR >110 ms but <120 ms is acceptable if there is no evidence of ventricular pre-excitation).
3. PR interval prolongation (>200 ms). Intermittent second (Type 1 second degree block [Wenckebach Phenomenon] while asleep is not exclusive]) or third degree atrioventricular (AV) block, or AV dissociation.
4. Persistent or intermittent complete bundle branch block (BBB), incomplete BBB, or intraventricular conduction delay with QRS >110 ms. Subjects with QRS >110 ms but <115 ms are acceptable if there is no evidence of eg, ventricular hypertrophy or pre-excitation.
5. Mean resting prolonged QTcF > 450 ms or shortened QTcF < 340 ms obtained from 3 ECGs.

10) A history of additional risk factors for torsades de pointes (TdP) (eg, chronic hypokalaemia not correctable with supplements, congenital or familial long QT syndrome, or family history of unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause TdP).

11) Known or suspected history of drug abuse, as judged by the PI. 12) Current smokers or those who have smoked or used nicotine products within the previous 30 days.

13) History of alcohol abuse or excessive intake of alcohol as judged by the PI.

14) Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate,) as judged by the PI.

15) Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of the IMP.

16) Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first admission on Study Day -1.

17) Use of any prescribed or non-prescribed medication including antacids, analgesics (other than use of ibuprofen) up to 72 hours before first dosing day until final follow-up visit, herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer (5 times half-life) if the medication has a long half-life.

18) Positive screen for drugs of abuse, cotinine (nicotine) and/or alcohol at screening or on each admission to the study centre .

19) History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to savolitinib or itraconazole.

20) Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.

21) Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days or 5 ½ lives (whichever is longer) of the first administration of IMP in this study.

Note: subjects consented and screened, but not randomized in this study or a previous Phase I study, are not excluded.

22) Involvement of any AstraZeneca, Parexel, or study centre employee or their close relatives 23) Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.

24) Subjects who are vegans, vegetarians or have medical dietary restrictions. 25) Subjects who cannot communicate reliably with the PI. 26) Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

27) Subjects who have previously received savolitinib.

In addition, any of the following is regarded as a criterion for exclusion from the genetic research:

28) Previous bone marrow transplant. 29) Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Savolitinib area under plasma concentration-time curve from time zero to infinity (AUC) ratios of geometric means of test treatment (savolitinib+itraconazole), relative to reference treatment (savolitinib alone) | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To assess the effect of itraconazole on the PK of savolitinib
Savolitinib maximum observed plasma concentration (Cmax) ratios of geometric means of test treatment (savolitinib+itraconazole), relative to reference treatment (savolitinib alone) | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To assess the effect of itraconazole on the PK of savolitinib

SECONDARY OUTCOMES:
Savolitinib:Area under the plasma concentration-curve from time zero to time of last quantifiable concentration [AUC(0-t)] ratios of geometric means of test treatment (savolitinib+itraconazole), relative to reference treatment (savolitinib alone) | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To assess the effect of itraconazole on the pharmacokinetics of metabolites M2 and M3
M2 and M3: Cmax ratios of geometric means of test treatment (savolitinib+itraconazole), relative to reference treatment (savolitinib alone) | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To assess the effect of itraconazole on the pharmacokinetics of metabolites M2 and M3
M2 and M3: AUC ratios of geometric means of test treatment (savolitinib+itraconazole), relative to reference treatment (savolitinib alone) | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To assess the effect of itraconazole on the pharmacokinetics of metabolites M2 and M3
M2 and M3: AUC(0-t) ratios of geometric means of test treatment (savolitinib+itraconazole), relative to reference treatment (savolitinib alone) | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To assess the effect of itraconazole on the pharmacokinetics of metabolites M2 and M3
Savolitinib, M2 and M3: Cmax | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Savolitinib, M2 and M3: AUC | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Savolitinib, M2 and M3: AUC(0-t) | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Savolitinib, M2 and M3: tmax | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Savolitinib, M2 and M3: t½,λz | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Savolitinib, M2 and M3: λz | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Savolitinib: CL/F | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Savolitinib: Vz/F | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Metabolite-to-parent ratios (MRCmax) | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Metabolite-to-parent ratios (MRAUC) | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Metabolite-to-parent ratios [MRAUC(0-t)] | Savolitinib,M2andM3:Treatment Periods1and3 (Study Days 1 and 18)pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose. Itraconazole:Treatment Period 3 (Study day 18)pre-dose, and 1 and 2 hours post-dose.
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with itraconazole
Number of subjects with adverse events | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in systolic blood pressure (BP) | Screening (Day -28), treatment period 1 (Study Day -1 and 1 to 14) and treatment period 3 (Study Day 1 to 3)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in diastolic BP | Screening (Day -28), treatment period 1 (Study Day -1 and 1 to 14) and treatment period 3 (Study Day 1 to 3)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in pulse rate | Screening (Day -28), treatment period 1 (Study Day -1 and 1 to 14) and treatment period 3 (Study Day 1 to 3)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in electrocardiogram (ECG) | Screening (Day -28), treatment period 1 (Days 1 to 14), treatment period 3 (Days 1 to 3) and follow-up visit (At least 14 days after last savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in physical examination | Study Day -1, Day 1 (pre-dose) of Treatment Periods 1, 2, and 3 (Study Days 1, 15, and 18)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in white blood cell (WBC) count | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in red blood cell (RBC) count | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in hemoglobin (Hb) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in hematocrit (HCT) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in mean corpuscular volume (MCV) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in mean corpuscular hemoglobin (MCH) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in mean corpuscular hemoglobin concentration (MCHC) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in neutrophils absolute count | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in lymphocytes absolute count | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in monocytes absolute count | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in eosinophils absolute count | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in basophils absolute count | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in platelets | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in reticulocytes absolute count | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in sodium | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in potassium | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in urea | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in creatinine clearence | Screening (Day -28 to Day -1)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in albumin | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in calcium | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in phosphate | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in glucose (fasting) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in C-reactive protein (CRP) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in alkaline phosphatase (ALP) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in alanine aminotransferase (ALT) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in aspartate aminotransferase (AST) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in gamma glutamyl transpeptidase (GGT) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in total bilirubin (TBL) | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in unconjugated bilirubin | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole
Number of subjects with abnormal findings in urinalysis | From Screening (Day -28) up to the Follow-up visit (at least 14 days after savolitinib dose)
  To assess the safety and tolerability of savolitinib in combination with itraconazole The parameters assessed will be glucose, protein and blood

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No